CLINICAL TRIAL: NCT03030963
Title: Effect of Equal Ratio Ventilation on Blood Loss During Posterior Lumbar Interbody Fusion Surgery: A Randomized Controlled Trial
Brief Title: Effect of Equal Ratio Ventilation on Blood Loss During Posterior Lumbar Interbody Fusion Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ji-young Kim, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3-2016-0241
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Blood Loss, Surgical
Keywords: Equal ratio ventilation(ERV); Peak inspiratory pressure(PIP); Blood loss; Posterior lumbar interbody fusion(PLIF); Prone position
MeSH Terms: conditions — Blood Loss, Surgical; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Equal-ratio ventilation(ERV) group (Experimental): ventilator inspiration to expiration ratio will be set 1:1.
  Interventions: Other: Equal ratio ventilation(ERV)
- Control group (Active Comparator): ventilator inspiration to expiration ratio will be set 1:2.
  Interventions: Other: I:E Ratio "1:2

INTERVENTIONS:
Other: Equal ratio ventilation(ERV) — Set the inspiratory to expiratory ratio 1:1 during mechanical ventilation
  Other Names: I:E ratio 1:1
  Arms: Equal-ratio ventilation(ERV) group
Other: I:E Ratio "1:2 — Set the inspiratory to expiratory ratio 1:2 during mechanical ventilation
  Arms: Control group

SUMMARY:
Ventilator mode change was associated with decrease in blood loss during posterior lumbar interbody fusion (PLIF) due to decrease in the peak inspiratory pressure (PIP). The purpose of this study was to determine the effect of equal ratio ventilation (ERV), which sets the I:E ratio of the ventilator to 1:1 during volume controlled ventilaiton, on surgical blood loss during PLIF. Investigators hypothesized that ERV would decrease surgical blood loss due to decrease in the PIP.

DETAILED DESCRIPTION:
After anesthesia, patients will receive ventilator settings according to theri group. The CVP will be measured before and after the prone position to ensure the proper positioning. Airway pressures including peak inspiratory pressure, mean/plateau airway pressure, arterial blood gas analysis data, hct, lactate, body temperature, mean arterial pressure, cardiac index. Recodings will be done 5min afte the induction, 5 min after the prone positioning, sikin suture, and 5min after supine position. Amount of bleeding, coagulation profile and Hct will be recorded 72 hrs after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age : 20~75 yr-old 2) Surgery : Posterior lumbar interbody fusion(PLIF) 2~3 levels

Exclusion Criteria:

* 1) Urgent or Emergency case 2) Previous lnstrumentation of lumbar spine (Exclusion : Discectomy, Partial hemilaminiectomy, etc) 3) Concurrent other operation 4) Patients who cannot understand informed consent (ex. Illiterate, Foreigner) 5) Obesity (BIM>30kg/m2) 6) Recent myocardial infarction (within 3 months) 7) Reduced left and right ventricular function (Ejection fraction<40%) or Congestive heart failure 8) Preoperative dysrhythmia 9) Aspirin or Plavix during perioperative periods 10) Lung disease 11) Chronic kidney disease or Dialysis 12) Severe hepatic disease

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03-04 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
The amount of intraoperative surgical bleeding | At the end of the surgery, approximately 4 hrs.
  The surgical blood loss was compared in the two groups (ERV vs. conrol) during posterior lumbar interbody fusion(PLIF) in prone position.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoung Kim, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No